CLINICAL TRIAL: NCT01106924
Title: Effects of Consumption of a Probiotic Formulation on Weight Control in Obese Subjects
Brief Title: Effects of a Probiotic on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08.22 NRC
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2011-09

CONDITIONS: Obesity
Keywords: Probiotics, Weight control, Body composition
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): daily probiotic consumption
  Interventions: Other: Probiotic
- Placebo (Placebo Comparator): daily placebo consumption
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic — daily probiotic consumption
  Arms: Probiotic
Other: Placebo — daily placebo consumption
  Arms: Placebo

SUMMARY:
Probiotics administration is associated with health benefits on gut barrier integrity and immunological functions of the gastrointestinal tract. Recently, probiotics consumption was proposed to reduce fat mass and body weight in rodents (Lee HY. et al. 2006; Hamad EM. et al. 2009) as well as abdominal fat in human (Kadooka Y, 2010). The mechanisms explaining the effects of probiotics in weight control are not well understood.

The primary objective of the clinical trial is to investigate whether a consumption of a probiotic formula when compared to an intake of a placebo, is associated with a greater reduction of body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 55 years old
* Weight: 30.0 kg/m2 ≤ BMI ≤ 39.9 kg/m2
* Non smokers
* Good general health
* A 2 weeks probiotics washout period prior to treatment initiation

Exclusion Criteria:

* Under antibiotics or treatments (medication or nutritional program) affecting body weight or glucose control for the last 3 months
* Currently participating or having participated in another clinical trial during the last 6 months prior to the beginning of this study
* Pregnant women, women who have given birth in the past year, women planning pregnancy in the next 6 months or menopausal women
* Excessive consumption of products enriched in probiotics (> 4 servings per week).
* History of drug or alcohol (> 2 drinks daily) abuse
* Abnormal thyroid hormone levels
* Intake of medication that could affect body weight and/or energy expenditure
* Family history of type 2 diabetes in first degree relatives
* Allergy to the ingredients in the study product and placebo
* Participant with anaemia
* Participant with a recent history of large weight fluctuations (e.g., > 10 kg in the past year
* Immune-compromised conditions
* Participant experiencing nausea, fever, vomiting, bloody diarrhoea or severe abdominal pain
* Participant with co-morbidity associated with obesity:

  * Hypertension (≥ 140/90 mm Hg)
  * Current use of antihypertensive medications, depression
  * Prediabetes (fasting glucose >100mg/dL)
  * Family history of premature coronary artery disease
  * LDL > 2.0 mmol/L
  * HDL < 1.3 mmol/L
  * Smoking
  * Obstructive sleep apnea
  * Type 2 diabetes
  * Cardiovascular disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Body weight; Body composition (DEXA); Waist circumference | PRE and POST

CONTACTS AND LOCATIONS:
Locations (1):
- Laval University and Laval Hospital, Québec, Quebec, Canada